CLINICAL TRIAL: NCT05735028
Title: A Preliminary Study on the Efficacy and Safety of PD-1/PD-L1 Inhibitors Combined With Centipeda Minima (CM) in Lung Cancer
Brief Title: The Efficacy and Safety of PD-1/PD-L1 Inhibitors Combined With Centipeda Minima (CM) in Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0826
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; Centipeda minima; efficacy; safty
MeSH Terms: conditions — Lung Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM group (Experimental): CM+PD-1/PD-L1 inhibitor
  Interventions: Drug: Centipeda minima+PD-1/PD-L1 inhibitor
- Control group (Active Comparator): PD-1/PD-L1 inhibitor
  Interventions: Drug: PD-1/PD-L1 inhibitor

INTERVENTIONS:
Drug: Centipeda minima+PD-1/PD-L1 inhibitor — Before routine anti-PD-1/PD-L1 treatment, patients were treated with Centipeda minima, and15g Centipeda minima decoction was taken twice a day for 5 consecutive days.
  Arms: CM group
Drug: PD-1/PD-L1 inhibitor — PD-1/PD-L1 inhibitor
  Arms: Control group

SUMMARY:
Lung cancer has a high global cancer morbidity and mortality. At present, PD-1/PD-L1 inhibitors have been approved by FDA to treat different types of lung cancer, but the efficacy is not good. There is an urgent need to develop drugs that can significantly enhance the efficacy of PD-1/PD-L1 inhibitors to enable tumor patients to obtain lasting anti-tumor response. Centipeda minima (CM), as a commonly used traditional Chinese medicine, is relatively safe. Previous studies found that it can inhibit the growth of lung cancer cells. At the level of animal research, the combined use of CM and PD-1/PD-L1 inhibitors produced a stronger anti-lung cancer effect, and did not produce obvious side effects on mice. Based on previous studies, the main purpose of this study was to evaluate the efficacy and safety of PD-1/PD-L inhibitors combined with herbivorous herbivores (CM) in the treatment of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-small cell lung cancer diagnosed by histopathology and intended to be treated with PD-1/PD-L1 inhibitors alone meet the following conditions:

1. Patients fully understand this study and voluntarily participate in and sign informed consent.
2. Patients with non-small cell lung cancer (NSCLC) confirmed by histopathology will be treated with PD-1/PD-L1 alone.
3. 18-70 years old, and the expected survival time is more than 6 months.
4. The indexes of stool routine are normal.

Exclusion Criteria:

1. Patients who plan to receive other traditional Chinese medicine treatment at the same time during the study period.
2. Those who are hypersensitive to any research drugs or ingredients
3. Those who have severe acute infection and are not controlled; or those who have suppurative and chronic infection and whose wounds are not healed.
4. Obvious gastrointestinal diseases during screening, such as inability to swallow, chronic diarrhea, intestinal obstruction, gastric ulcer and so on.
5. Those who have participated in clinical trials of other drugs within 5 or 4 weeks.
6. Patients with severe heart disease, including congestive heart failure, uncontrollable high-risk arrhythmias, unstable angina pectoris, myocardial infarction, severe valvular heart disease and intractable hypertension.
7. Suffering from uncontrollable neurological, mental illness or mental disorders, poor compliance, unable to cooperate and describe the treatment response. Primary brain tumor or central nervous system metastasis is not controlled, with obvious intracranial hypertension or neuropsychiatric symptoms.
8. Those with bleeding tendency; evidence of hereditary hemorrhagic physique or blood coagulation disorder
9. Severe allergic / allergic reaction to humanized antibody.
10. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days prior to the first administration of the study, allowing the use of physiological doses of glucocorticoids (prednisone or equivalent for ≤ 10mg/ days).
11. Exclude subjects with active, known or suspected autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hypothyroidism, including but not limited to these diseases or syndromes).
12. Vulnerable groups: such as patients with serious diseases, incapacitated, illiterate, mentally retarded / related mental disorders, children.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion, an average of 2 year.
  Progression-free survival
the temperature | through study completion, an average of 2 year.
  Vital signs
blood pressure | through study completion, an average of 2 year.
  Vital signs
complete blood count | through study completion, an average of 2 year.
  laboratory index
adverse event and severe adverse event | through study completion, an average of 2 year.
  adverse event and severe adverse event, according to NCI-CTC V5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 2 year.
  Objective Response Rate
disease control rate (DCR) | through study completion, an average of 2 year.
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Ying Dong, Doctorate, Principal Investigator — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No